CLINICAL TRIAL: NCT04456946
Title: Prospective Investigation of the Effects of Different Treatment Techniques on Myofascial Trigger Points in Patients With Temporomandibular Dysfunction (TMD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ahmet Faruk ERTURK, Lecturer, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/72; 34978 (Other Grant/Funding Number: Scientific Research Projects Coordination Unit of Istanbul University); 2019-190 (Other: Republic of Turkey Ministry of Health)
Record Dates: First submitted 2020-06-23; First posted 2020-07-07 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Low Level Laser and Occlusal Splint
Keywords: Low Level Laser; Occlusal Splint; Temporomandibular Disfunction
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of Low Level Laser Therapy (Experimental)
  Interventions: Device: Low Level Laser Therapy
- Group of Occlusal Splint Treatment (Experimental)
  Interventions: Device: Occlusal Splint Treatment

INTERVENTIONS:
Device: Low Level Laser Therapy — Low Level Laser Therapy
  Arms: Group of Low Level Laser Therapy
Device: Occlusal Splint Treatment — Occlusal Splint Treatment
  Arms: Group of Occlusal Splint Treatment

SUMMARY:
In the literature, there are no studies comparing the use of occlusal splint and Low Level Laser (LLL) in the treatment of Temporomandibular Disfunction (TMD) and including Ultrasonography (USG) in these parameters. In this study, it is aimed to contribute to the literature in terms of determining which treatment method is more effective by evaluating the changes in the needles muscles with the use of occlusal splints and LLL with USG and other parameters in certain periods, as well as evaluating which parameters are more effective.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 who apply with Temporomandibular Joint (TMJ) problems
* Patients with pain in the joint and chewing muscle area

Exclusion Criteria:

* Syndromic patients
* Patients under the age of 18
* Patients with a history of orthognathic surgery
* Pregnants
* Antidepressant Users
* Patients Using Removable Dentures
* Patients who have had joint treatment in the past six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Joint Pain Scale | 2 years
  Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD) form will be used in our study

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Faruk Erturk, Assistant Professor, Principal Investigator — Biruni University
Locations (1):
- Istanbul University, Dentistry Faculty, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/46/NCT04456946/Prot_SAP_001.pdf
  • Informed Consent Form (2019-09-12): https://cdn.clinicaltrials.gov/large-docs/46/NCT04456946/ICF_000.pdf